CLINICAL TRIAL: NCT03291496
Title: Microfluidic Assessment of Clinical Outcomes in Preterm Newborns
Status: Active, not recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201701566 N; R01HD089939 (NIH); OCR26202 (Other: OCR OnCore)
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Neonatal SEPSIS
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Preterm Neonates: Blood collection Preterm. From blood, the speed, directionality, and persistence of PMN chemotaxis using microfluidic devices and transcriptomic analysis will be measured.
  Interventions: Other: Blood Collection Preterm
- Term Neonates: Blood collection Term. From blood, the speed, directionality, and persistence of PMN chemotaxis using microfluidic devices and transcriptomic analysis will be measured.
  Interventions: Other: Blood Collection Term
- Healthy Adult: One-time whole blood draw of 1ml collection
  Interventions: Other: Adult Blood collection

INTERVENTIONS:
Other: Blood Collection Preterm — Blood will be collected on day 4 of life and then approximately every 3 days until 21 days of life. Thereafter, one sample will be collected weekly until discharge. For preterm neonates that have suspected sepsis an additional sample will be collected within 24-48 hours of the initial sepsis evaluation.
  Groups: Preterm Neonates
Other: Blood Collection Term — A single 250 µl blood sample will be collected once the term neonate is >24 hours old.
  Groups: Term Neonates
Other: Adult Blood collection — One Time 1 ml of whole blood collected
  Groups: Healthy Adult

SUMMARY:
Sepsis has its greatest impact in the prematurely born (preterm) population. Neonatal sepsis (sepsis within the first month of life) causes over one million deaths worldwide annually, and is one of the most common, difficult and costly problems to diagnose, treat and prevent. The preterm infant can suffer rates of sepsis up to 1000-fold higher than the full-term infant, and bears the brunt of the associated mortality and lifelong sepsis-survivor morbidity.

The project is enabled by several novel, validated, microfluidic technologies that are robust and easy to use with little training. These technologies provide comprehensive measures of the functionality of blood PMN population; a critical cellular component of innate immunity. The study team will also extract high-quality nucleic acids from microfluidic-sorted PMNs for transcriptomic analyses. Collectively, these techniques require a total of 250 microliters (µL) of blood, which makes them particularly useful for preterm infants where sample volume is limited, and facilitates serial assessments with unprecedented temporal resolution of key functions of PMNs.

These studies, integrated with bioinformatics approaches, will generate new tools for diagnosing sepsis in the newborn and predicting clinical outcomes. Such approaches have the capability to dramatically change the clinical management of the preterm infant, and potentially improve long-term outcomes while reducing hospital costs.

DETAILED DESCRIPTION:
Blood samples will be collected from two populations: preterm infants and term infants.

1. Preterm neonates (<32 weeks) the study team will collect a baseline 250 µl blood sample on day four of life and then approximately every three days, as is possible, until twenty-one days of life. In addition, for preterm neonates who have suspected sepsis, an additional 250 µl blood sample will be obtained on the day of suspected sepsis. After day twenty-one of life, 250 µl blood will be sampled one time per week until discharge, when a final 250 µl blood sample will be collected. The amount drawn for study related blood collections will not exceed the lesser of 50 ml or 3.0 ml/kg in an 8-week period.
2. Term neonates (>36 weeks) the study team will be collect a single 250 µl blood sample with the routine screen for metabolic disorders when they are >24 hours old. This will be the only study related blood collection for term neonates.

For all infants, term and preterm, the following data will be collected while the neonate is hospitalized: Demographic information (age, date of birth), past and present medical records, laboratory, microbiology, and all other test results, X-ray, CT, MRI, US and all other imaging test results, records about any medication received during admission, records of physical exam during admission, records of all vital signs and hemodynamic monitoring during admission, records of any procedure or intervention during admission, and condition at the discharge and discharge location.

ELIGIBILITY:
Inclusion Criteria:

* For preterm neonates <32 weeks gestation at birth with no known or suspected congenital anomalies.
* For term neonates >36 weeks gestation at birth with no known or suspected congenital anomalies.

Exclusion Criteria:

* Congenital defects, suspected genetic disorders, 32-36 weeks completed gestation, or lack of consent.

Healthy Adult:

* Inclusion criteria Between the ages of 18 and 65 years of age
* Exclusion Criteria Taking any immune modifying medications or have an active immune modifying disease process

Ages: 23 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm neonates <32 weeks gestation. Term neonates >36 weeks gestation.
Sampling Method: Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of Sepsis in Premature Neonates | Days 4-21
  The study team will determine whether blood neutrophil migration phenotype using a microfluidic-based approach can be used to predict the onset of sepsis, as well as poor outcome from sepsis, in premature neonates. From peripheral blood, the study team will measure speed, directionality, and persistence of neutrophil chemotaxis using microfluidic devices. The goal is to prospectively identify and validate biomarkers that can stratify neonates who will become septic and have a protracted clinical course. To complement these functional assays, the study team will determine if transcriptomic profiling adds to the diagnostic resolution generated through these functional analyses.

SECONDARY OUTCOMES:
Neutrophil Function of Premature Neonate during Development | Days 22-180
  The study team will determine whether premature neonates restore a more normal neutrophil migration phenotype and genomic profile as they reach their developmental milestones during NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: James L Wynn, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu L, Johnson HL, Cousens S, Perin J, Scott S, Lawn JE, Rudan I, Campbell H, Cibulskis R, Li M, Mathers C, Black RE; Child Health Epidemiology Reference Group of WHO and UNICEF. Global, regional, and national causes of child mortality: an updated systematic analysis for 2010 with time trends since 2000. Lancet. 2012 Jun 9;379(9832):2151-61. doi: 10.1016/S0140-6736(12)60560-1. Epub 2012 May 11. PMID 22579125
- [Background] INIS Collaborative Group; Brocklehurst P, Farrell B, King A, Juszczak E, Darlow B, Haque K, Salt A, Stenson B, Tarnow-Mordi W. Treatment of neonatal sepsis with intravenous immune globulin. N Engl J Med. 2011 Sep 29;365(13):1201-11. doi: 10.1056/NEJMoa1100441. PMID 21962214
- [Background] Barton L, Hodgman JE, Pavlova Z. Causes of death in the extremely low birth weight infant. Pediatrics. 1999 Feb;103(2):446-51. doi: 10.1542/peds.103.2.446. PMID 9925839
- [Background] Stoll BJ, Hansen NI, Bell EF, Shankaran S, Laptook AR, Walsh MC, Hale EC, Newman NS, Schibler K, Carlo WA, Kennedy KA, Poindexter BB, Finer NN, Ehrenkranz RA, Duara S, Sanchez PJ, O'Shea TM, Goldberg RN, Van Meurs KP, Faix RG, Phelps DL, Frantz ID 3rd, Watterberg KL, Saha S, Das A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal outcomes of extremely preterm infants from the NICHD Neonatal Research Network. Pediatrics. 2010 Sep;126(3):443-56. doi: 10.1542/peds.2009-2959. Epub 2010 Aug 23. PMID 20732945
- [Background] Martin GS, Mannino DM, Moss M. The effect of age on the development and outcome of adult sepsis. Crit Care Med. 2006 Jan;34(1):15-21. doi: 10.1097/01.ccm.0000194535.82812.ba. PMID 16374151
- [Background] Cohen-Wolkowiez M, Moran C, Benjamin DK, Cotten CM, Clark RH, Benjamin DK Jr, Smith PB. Early and late onset sepsis in late preterm infants. Pediatr Infect Dis J. 2009 Dec;28(12):1052-6. doi: 10.1097/inf.0b013e3181acf6bd. PMID 19953725
- [Background] Watson RS, Carcillo JA. Scope and epidemiology of pediatric sepsis. Pediatr Crit Care Med. 2005 May;6(3 Suppl):S3-5. doi: 10.1097/01.PCC.0000161289.22464.C3. PMID 15857554
- [Background] Girard TD, Opal SM, Ely EW. Insights into severe sepsis in older patients: from epidemiology to evidence-based management. Clin Infect Dis. 2005 Mar 1;40(5):719-27. doi: 10.1086/427876. Epub 2005 Jan 28. PMID 15714419
- [Background] Haque KN, Khan MA, Kerry S, Stephenson J, Woods G. Pattern of culture-proven neonatal sepsis in a district general hospital in the United Kingdom. Infect Control Hosp Epidemiol. 2004 Sep;25(9):759-64. doi: 10.1086/502473. PMID 15484801
- [Background] Martinot A, Leclerc F, Cremer R, Leteurtre S, Fourier C, Hue V. Sepsis in neonates and children: definitions, epidemiology, and outcome. Pediatr Emerg Care. 1997 Aug;13(4):277-81. doi: 10.1097/00006565-199708000-00011. No abstract available. PMID 9291519
- [Background] Stoll BJ, Hansen NI, Adams-Chapman I, Fanaroff AA, Hintz SR, Vohr B, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental and growth impairment among extremely low-birth-weight infants with neonatal infection. JAMA. 2004 Nov 17;292(19):2357-65. doi: 10.1001/jama.292.19.2357. PMID 15547163
- [Background] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. Changes in pathogens causing early-onset sepsis in very-low-birth-weight infants. N Engl J Med. 2002 Jul 25;347(4):240-7. doi: 10.1056/NEJMoa012657. PMID 12140299
- [Background] Stoll BJ, Hansen N, Fanaroff AA, Wright LL, Carlo WA, Ehrenkranz RA, Lemons JA, Donovan EF, Stark AR, Tyson JE, Oh W, Bauer CR, Korones SB, Shankaran S, Laptook AR, Stevenson DK, Papile LA, Poole WK. Late-onset sepsis in very low birth weight neonates: the experience of the NICHD Neonatal Research Network. Pediatrics. 2002 Aug;110(2 Pt 1):285-91. doi: 10.1542/peds.110.2.285. PMID 12165580
- [Background] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Background] Clark RH, Bloom BT, Spitzer AR, Gerstmann DR. Reported medication use in the neonatal intensive care unit: data from a large national data set. Pediatrics. 2006 Jun;117(6):1979-87. doi: 10.1542/peds.2005-1707. PMID 16740839
- [Background] Bizzarro MJ, Dembry LM, Baltimore RS, Gallagher PG. Changing patterns in neonatal Escherichia coli sepsis and ampicillin resistance in the era of intrapartum antibiotic prophylaxis. Pediatrics. 2008 Apr;121(4):689-96. doi: 10.1542/peds.2007-2171. PMID 18381532
- [Background] Hill DA, Hoffmann C, Abt MC, Du Y, Kobuley D, Kirn TJ, Bushman FD, Artis D. Metagenomic analyses reveal antibiotic-induced temporal and spatial changes in intestinal microbiota with associated alterations in immune cell homeostasis. Mucosal Immunol. 2010 Mar;3(2):148-58. doi: 10.1038/mi.2009.132. Epub 2009 Nov 25. PMID 19940845
- [Background] Jernberg C, Lofmark S, Edlund C, Jansson JK. Long-term impacts of antibiotic exposure on the human intestinal microbiota. Microbiology (Reading). 2010 Nov;156(Pt 11):3216-3223. doi: 10.1099/mic.0.040618-0. Epub 2010 Aug 12. PMID 20705661
- [Background] Cotten CM, Taylor S, Stoll B, Goldberg RN, Hansen NI, Sanchez PJ, Ambalavanan N, Benjamin DK Jr; NICHD Neonatal Research Network. Prolonged duration of initial empirical antibiotic treatment is associated with increased rates of necrotizing enterocolitis and death for extremely low birth weight infants. Pediatrics. 2009 Jan;123(1):58-66. doi: 10.1542/peds.2007-3423. PMID 19117861
- [Background] Sjogren YM, Tomicic S, Lundberg A, Bottcher MF, Bjorksten B, Sverremark-Ekstrom E, Jenmalm MC. Influence of early gut microbiota on the maturation of childhood mucosal and systemic immune responses. Clin Exp Allergy. 2009 Dec;39(12):1842-51. doi: 10.1111/j.1365-2222.2009.03326.x. Epub 2009 Sep 3. PMID 19735274
- [Background] Wynn JL, Neu J, Moldawer LL, Levy O. Potential of immunomodulatory agents for prevention and treatment of neonatal sepsis. J Perinatol. 2009 Feb;29(2):79-88. doi: 10.1038/jp.2008.132. Epub 2008 Sep 4. PMID 18769381
- [Background] Wynn J, Cornell TT, Wong HR, Shanley TP, Wheeler DS. The host response to sepsis and developmental impact. Pediatrics. 2010 May;125(5):1031-41. doi: 10.1542/peds.2009-3301. Epub 2010 Apr 26. PMID 20421258
- [Background] Strunk T, Currie A, Richmond P, Simmer K, Burgner D. Innate immunity in human newborn infants: prematurity means more than immaturity. J Matern Fetal Neonatal Med. 2011 Jan;24(1):25-31. doi: 10.3109/14767058.2010.482605. Epub 2010 Jun 23. PMID 20569168
- [Background] Wynn JL, Scumpia PO, Winfield RD, Delano MJ, Kelly-Scumpia K, Barker T, Ungaro R, Levy O, Moldawer LL. Defective innate immunity predisposes murine neonates to poor sepsis outcome but is reversed by TLR agonists. Blood. 2008 Sep 1;112(5):1750-8. doi: 10.1182/blood-2008-01-130500. Epub 2008 Jun 30. PMID 18591384
- [Background] Wynn JL, Scumpia PO, Delano MJ, O'Malley KA, Ungaro R, Abouhamze A, Moldawer LL. Increased mortality and altered immunity in neonatal sepsis produced by generalized peritonitis. Shock. 2007 Dec;28(6):675-683. doi: 10.1097/SHK.0b013e3180556d09. PMID 17621256
- [Background] PrabhuDas M, Adkins B, Gans H, King C, Levy O, Ramilo O, Siegrist CA. Challenges in infant immunity: implications for responses to infection and vaccines. Nat Immunol. 2011 Mar;12(3):189-94. doi: 10.1038/ni0311-189. No abstract available. PMID 21321588
- [Background] Wynn JL, Cvijanovich NZ, Allen GL, Thomas NJ, Freishtat RJ, Anas N, Meyer K, Checchia PA, Lin R, Shanley TP, Bigham MT, Banschbach S, Beckman E, Wong HR. The influence of developmental age on the early transcriptomic response of children with septic shock. Mol Med. 2011;17(11-12):1146-56. doi: 10.2119/molmed.2011.00169. Epub 2011 Jul 5. PMID 21738952
- [Background] Goldstein B, Giroir B, Randolph A; International Consensus Conference on Pediatric Sepsis. International pediatric sepsis consensus conference: definitions for sepsis and organ dysfunction in pediatrics. Pediatr Crit Care Med. 2005 Jan;6(1):2-8. doi: 10.1097/01.PCC.0000149131.72248.E6. PMID 15636651
- [Background] Wynn JL, Guthrie SO, Wong HR, Lahni P, Ungaro R, Lopez MC, Baker HV, Moldawer LL. Postnatal Age Is a Critical Determinant of the Neonatal Host Response to Sepsis. Mol Med. 2015 Jun 2;21(1):496-504. doi: 10.2119/molmed.2015.00064. PMID 26052715
- [Background] Nathan C. Neutrophils and immunity: challenges and opportunities. Nat Rev Immunol. 2006 Mar;6(3):173-82. doi: 10.1038/nri1785. PMID 16498448
- [Background] Squire E, Favara B, Todd J. Diagnosis of neonatal bacterial infection: hematologic and pathologic findings in fatal and nonfatal cases. Pediatrics. 1979 Jul;64(1):60-4. PMID 450562
- [Background] Wong HR, Freishtat RJ, Monaco M, Odoms K, Shanley TP. Leukocyte subset-derived genomewide expression profiles in pediatric septic shock. Pediatr Crit Care Med. 2010 May;11(3):349-55. doi: 10.1097/PCC.0b013e3181c519b4. PMID 20009785
- [Background] Wynn JL, Wong HR. Pathophysiology and treatment of septic shock in neonates. Clin Perinatol. 2010 Jun;37(2):439-79. doi: 10.1016/j.clp.2010.04.002. PMID 20569817